CLINICAL TRIAL: NCT04141163
Title: A Parallel Group Design Randomized Double-Blind Trial of Metformin Treatment in Patients With Fragile X Syndrome on Safety and Effects on Cognition, Anxiety, Attention and Biomarkers
Brief Title: Metformin in Patients With Fragile X
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rowan University (Other)
Collaborators: FRAXA Research Foundation (Other); University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Sean McBride, M.D., Ph.D., Associate Professor, Rowan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro2018000310
Record Dates: First submitted 2019-10-24; First posted 2019-10-28 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Metformin (Experimental): Subjects randomized to metformin will start at 500mg once a day for 7 days and increase as is tolerated to 500mg twice a day for 7 days, then to 1000mg in the morning and 500mg at dinner for 7 days and then to the target dose of 1,000mg twice a day.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Subjects randomized to placebo will start at 500mg once a day for 7 days and increase as is tolerated to 500mg twice a day for 7 days, then to 1000mg in the morning and 500mg at dinner for 7 days and then to the target dose of 1,000mg twice a day.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Metformin — Metformin, 1,1 dimethylbiguanide, or systematic (IUPAC) name N,N-dimethylimidodicarbonimidic diamide, is an oral anti-diabetic medicine approved in the US by the FDA in 1994. It is marketed alone under the names metformin (generic), Glucophage XR, Riomet, Fortamet, Glumetza, Obimet, Gluformin, Dianben, Diabex, and Diaformin and in combination with other drugs under the names Actoplus Met, Metaglip, Glucovance, Janumet, Kombiglyze XR, and PrandiMet
  Other Names: glucophage
  Arms: Metformin
Drug: Placebo oral tablet — No therapeutic effect
  Arms: Placebo

SUMMARY:
The purpose of this trial is to investigate the use of metformin in the treatment of Fragile X syndrome (FXS) patients. Metformin is an FDA approved compound with an established safety profile and minimal side effects that specifically targets and normalizes multiple aspects of the pathophysiology in FXS. This is a randomized double-blind placebo-controlled 2-arm parallel group design study of the drug metformin and placebo in FXS subjects with a primary outcome measure of safety/tolerability and secondary outcome measures on cognition, attention, anxiety, sleep, and physiologic and biochemical biomarkers.

DETAILED DESCRIPTION:
This trial will be a randomized placebo controlled, double-blind, parallel group design study of treatment with metformin on the primary outcome of safety/tolerance with secondary outcome measurements of the effects on cognition (encompassing social and repetitive behavior), attention, anxiety, and physiological and biochemical biomarkers of patients with FXS. FXS represents a well-defined population of ASD in which to test a specific targeted treatment looking at a well-defined set of cognitive and bioassay measures.

Trial length is designed to have a chance at seeing if the medication can improve cognitive outcome measures. The study duration includes the screening period and a 24-week single-blind drug/placebo phase.

ELIGIBILITY:
Inclusion Criteria:

* Male between the ages of 16-50 years old at the time of consent
* Diagnosis of full mutation FXS.
* Stable on any psychoactive medication for at least 4 weeks before receiving study drug, including antidepressants, stimulants, antipsychotics, and mood stabilizers.
* Seizure free for at least the past 3 months.
* No major health issues or diseases expected to interfere with the study
* No history of diabetes
* Not currently taking metformin at the time of enrollment
* Average basal blood glucose HgbA1c < 7.0
* Study partner with frequent contact with patient willing to accompany patient to visits and complete caretaker/partner study forms
* No contraindication to metformin
* Willing to complete all baseline assessments and study procedures

Exclusion Criteria:

* Has a medical condition that would make treatment unsafe such as diabetes, pancreatic disease, liver or kidney disease, a history of epilepsy or seizure disorder that is not controlled, as well as any other medical condition as determined by the study doctor.
* Has an eating disorder that has been clinically diagnosed, predisposing them to low BMI.
* Has received any investigational compound within 30 days prior to the first dose of study medication.
* Has received metformin in a previous clinical study or as a therapeutic agent.
* Is an immediate family member, study site employee, or in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling), or may consent under duress.
* Has uncontrolled, clinically significant neurological, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, or endocrine disease or other abnormality which may impact the ability of the participant to participate or potentially confound the study results.
* Has a known hypersensitivity to any component of the formulation of metformin.
* Has a history of drug abuse (defined as any illicit drug use) or a history of alcohol abuse within 6 months prior to the screening visit or is unwilling to agree to abstain from alcohol and drugs throughout the study.
* Currently taking any excluded medication, supplements, or food products, or has taken any in the 3 weeks preceding Visit 1. This includes carbonic anhydrase inhibitors and the medication topamax.
* Has evidence of current cardiovascular, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma hypoxemia, hypertension or allergic skin rash. There is any finding in the participant's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking metformin or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to uncontrolled seizure disorders, and cardiac arrhythmias.
* History of any surgical intervention known to impact absorption (e.g., bariatric surgery or bowel resection).
* Compromised renal function at screening as determined by creatinine levels >1.5mg/dL and/or creatinine clearance <45mL/min based on Cockcroft-Gault calculation.
* Liver dysfunction at screening as evidenced by alanine transaminase (ALT/SGPT) values > 2X upper limit of normal or aspartate transaminase (AST/SGOT) values > 3X upper limit of normal or total bilirubin > 2X upper limit of normal.
* Has donated or lost 450 mL or more of his blood volume (including plasmapheresis), or had a transfusion of any blood product within 3 months prior to Day 1.
* Has a history of abnormal (clinically significant) electrocardiogram (ECG). Entry of any participant with an abnormal (not clinically significant) ECG must be approved, and documented by signature by the principal investigator.
* Has abnormal Screening or Day 1 vital sign values that suggest a clinically significant underlying disease.
* Is at risk of suicide, has made a suicide attempt within the last year or has current active suicidal ideation. In accordance with previous FDA regulated studies on patients with FXS this determination will include asking 3 questions. 1) Has the subject made a suicide attempt? 2) Has the subject expressed any (active) suicidal thoughts or intent to harm him/herself or others? 3) Has there been a significant increase in the severity or frequency of self-injurious behaviors, or harm toward others, such that continued safety is a concern?
* Laboratory abnormalities in B12, or other common lab parameters that might contribute to cognition or participation in study
* In the opinion of the investigator or sponsor, the participant is unsuitable for inclusion in the study.

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-10-29 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
The safety and tolerability of metformin in patients with Fragile X Syndrome as assessed by the number of adverse events reported during the course of the study. | 1-2 years
  measured by the number of reported adverse events, assessed using the Safety Monitoring Uniform Report Form (SMURF), modified for metformin use

SECONDARY OUTCOMES:
Patients taking Metforming have improved cognition, sleep, attention or anxiety from baseline to the end of the study | 1-2 years
  measured by a variety of questionnaires and assessments done throughout the length of the study

CONTACTS AND LOCATIONS:
Overall Officials: Sean McBride, MD, PhD, Principal Investigator — Rowan University
Locations (1):
- Rowan University School of Osteopathic Medicine, Stratford, New Jersey, United States